CLINICAL TRIAL: NCT04224870
Title: A Single Cohort Study Collecting Interval Timed Incisional Epidermal and Dermal Tissue Samples During Surgical Procedures to Profile Temporal Response of Tissue After Noxious Stimuli.
Brief Title: Collecting Interval Timed Incisional Epidermal and Dermal Tissue Samples During Surgical Procedures to Profile Temporal Response of Tissue After Noxious Stimuli
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 200031; 20-CC-0031
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04-17

CONDITIONS: Abdominal Surgery; Thoracic Surgery; Urological Surgery
Keywords: Epidermal; Transcriptomics; Dermal; Surgery; Incision; Natural History
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical Incision: A single cohort study, of 12 participants with a scheduled surgical procedure, of at least 4 hours, for up to six (6) timed tissue sampling at surgical incision. No investigational therapy is planned.

SUMMARY:
Background:

Opioids are a class of drug that are often used to manage pain after a person has surgery. Because of the current opioid crisis, researchers want to improve ways to manage pain after surgery with fewer side effects. To do this, they need to understand pain better. In this study, they want to measure chemical reactions and find genes involved in producing the pain that people feel after surgery.

Objective:

To find the pain signals starting at the site of skin incision during surgery.

Eligibility:

People age 18 and older who are having a surgery that will last for at least 4 hours.

Design:

The participant s primary surgeon will make sure he or she is eligible for surgery.

Participants will complete a generalized pain questionnaire before the day of surgery. This will give a baseline measurement.

During surgery, 4 to 6 tissue samples at the site of incision will be taken at the following time points:

when the surgery starts

at 1, 2, 4, and 6 hours

when the wound is closed (if the surgery lasts longer than 8 hours).

The samples will only be taken if they will not prevent the wound from healing properly.

For the first 2 days after surgery, participants will complete short questionnaires about their level of pain. Each will take less than 5 minutes to complete. Their answers will be protected....

DETAILED DESCRIPTION:
Background:

* Opioids are the cornerstone of postoperative pain management. However, in light of the current opioid crisis, there is a recognized need for improved postoperative pain management to address pain with fewer side effects.
* New pain medications that are as effective and less problematic are a goal but much of the foundational knowledge required to meet these need is underdeveloped in human studies and are derived from rodent studies.
* We propose to identify critical human tissue nociceptive signals originating at the site of surgical incision initiating the pain response to identify biomarkers of human cutaneous pain signaling.
* Mechanisms of pain and pain sensitivities originating at the surgical site are not well understood.
* Clinical and basic research can unlock the etiology of surgical incisional pain and direct biomedicine to better address this area of underdeveloped research both now and in the future; uniquely providing opportunities to perform important studies on gene expression.

Objectives:

* Identification of transcriptional alterations in epidermal and dermal tissue of at least four (4), but up to six (6) time points during surgical procedures.
* Tandem mass spectrometry (MS/MS) measurement from human epidermal sample to identify alterations in candidate oxylipins and peptide mediators of pain, inflammation and itch.

Eligibility:

-Male or female, aged 18 years and older that are consented for a primary surgical procedure of greater than four (4) hours. Participants without skin abnormalities at tissue sampling site.

Design:

-A single cohort study, of 12 surgical participants with a scheduled surgical procedure, of at least 4 hours, at the NIH Clinical Center, for up to six (6) timed tissue sampling at surgical incision. No investigational therapy is planned.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Male or female, aged 18 years and older. Participant will be consented for a surgical procedure (primary surgical protocol) anticipated to last longer than 4 hours.
2. Cutaneous incisional tissue sample (removal) is determined by surgeon not to compromise the incisional closure.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Participants with known skin abnormalities (dermatologic /dermatitis conditions): psoriasis, atopic dermatitis, rosacea, cancer melanomas, basal cell as well as benign lesions, tissue burns, infections, hematomas, and contusions) at the surgical site.
2. Participants with pre-existing scar tissue at the incision site and/or a history of surgical procedures at the same site. Pre-existing scar tissue will confound the results since the baseline is different from normal non-scar tissue and therefore cannot be used as a basis for comparison.
3. Participants with a history of radiation treatment at the incision site, when the incision site was included in the radiation field.
4. Participants with other skin conditions that would compromise epidermal and dermal samples in the opinion of the surgeon.
5. Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations (within 6 months) that would limit compliance with study requirements.
6. The pain questionnaire will be only available in English, therefore non-English speaking/reading participants are excluded from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a tissue procurement research protocol, recruiting twelve (12) adult participants for incision tissue procurement during surgical procedures greater than four (4) hours. Potential participants are surgical candidates referred from various surgical services within the Clinical Research Center (CRC); evaluation and interest in this study will be facilitated by the primary surgeon. Once primary informed consent is obtained, the potential participant will be approached by our research team to discuss the tissue procurement study in further detail, and if interested, will be given a Read Only informed consent document to review. On preoperative admission to the CRC, research team members identified in the protocol as able to obtain consent will visit the participant and review the study. Interested participants will formally sign study consent at this time.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-11-07 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Quantitative measurements | end of study
  Quantitative measurements of all expressed transcripts (by RNA-Seq) at each time point collected during surgery (initial incision, 1h, 2h, 4h, 6h, and closure). This will identify the most notable genes according to significance, expression level and fold-change.

SECONDARY OUTCOMES:
Tandem mass spectrometry (MS/MS) | end of study
  The endpoint of MS/MS is a quantitative estimate of abundance of the examined molecule (oxylipin or peptide mediators).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Mannes, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-CC-0031.html